CLINICAL TRIAL: NCT04764318
Title: A Pilot Study of Hypertension Management Using Remote Patient Monitoring: Study 2
Brief Title: Hypertension Management Using Remote Patient Monitoring: Study 2
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Omron Healthcare Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Stephen Persell, MD, MPH, Professor of Medicine, Northwestern University
Other Study IDs: STU00213093 Study 2
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Remote Patient Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Remote patient monitoring for hypertension: All intervention practices will receive communication by email explaining RPM procedures, ordering, use, and financial implications. We will also present this information at practice meetings. Primary care clinicians at these sites will receive clinical decision support (Epic Best Practice Alert) for patients meeting primary or secondary eligibility criteria. It will be at the discretion of the primary care clinicians when to offer or refer patients to RPM.
  Interventions: Behavioral: Remote patient monitoring for hypertension
- Remote patient monitoring with care management: All intervention practices will receive communication by email explaining RPM procedures, ordering, use, and financial implications. We will also present this information at practice meetings. Primary care clinicians at these sites will receive clinical decision support (Epic Best Practice Alert) for patients meeting primary or secondary eligibility criteria. It will be at the discretion of the primary care clinicians when to offer or refer patients to RPM. In addition, PCPs will receive lists of candidate patients. Care managers will assist with the outreach to patients to offer RPM when recommended by the PCP, will monitor and support patient use of the remote monitor, and will promote action on the part of the patient or PCP when uncontrolled hypertension is present.
  Interventions: Behavioral: Remote patient monitoring with care management
- Usual care: Medicare patients from non-intervention primary care practices in Northwestern Medical Group will contribute EHR data but will not have any new procedures put in place.

INTERVENTIONS:
Behavioral: Remote patient monitoring for hypertension — The intervention involves making available remote physiologic monitoring services for hypertension patients allowable under Medicare for blood pressure (and weight if desired) when ordered by a patient's clinician.
  Groups: Remote patient monitoring for hypertension
Behavioral: Remote patient monitoring with care management — The intervention involves making available remote physiologic monitoring services for hypertension patients allowable under Medicare for blood pressure (and weight if desired) when ordered by a patient's clinician and providing care management services to support the enrollment and active use of this service.
  Groups: Remote patient monitoring with care management

SUMMARY:
The investigators will conduct a pragmatic pilot test of a remote patient monitoring system (RPM) for blood pressure measurement for Medicare patients with hypertension with and without the support of a care management program. The primary objective is to better understand how patients' remote monitoring of blood pressure and the direct transmission of this data to a healthcare system's EHR can be used by the patient and the care team to support optimal hypertension care and whether the addition of active care management increases the use of RPM and improvements in blood pressure.

This pilot study will be conducted in four Northwestern Medical Group (NMG) primary care practices. Two practices will have RPM available for primary care physicians to order for their eligible Medicare patients and two practices will also receive the support of a care management program to assist with patient enrollment, blood pressure monitoring and taking action in the setting of uncontrolled blood pressure.

The investigators will conduct a pragmatic non-blinded, non-randomized pilot study with contemporaneous controls among NMG outpatient clinics that provide adult primary care. They will make comparisons of data obtained through the course of routine care delivery from pilot and non-pilot practices.

ELIGIBILITY:
Inclusion Criteria:We will use these criteria to determine which patients will be included or excluded in the study analytic data set.

General inclusion criteria:

* Adults aged 65 to 85 years at the time of the study start date
* Receive their primary care from an eligible Northwestern Medicine clinic site
* One or more office or telehealth visits in the year preceding the study start date

Inclusion criteria primary population:

* Last two office blood pressures ≥140 mm Hg systolic or ≥90 mmHg diastolic
* Diagnosis of hypertension in the year preceding the study start date (problem list or encounter diagnosis)

Inclusion criteria for secondary population

* Meet criteria for primary population OR
* Diagnosed hypertension but did not have the last two office blood pressures ≥140 mm Hg systolic or ≥90 mmHg diastolic OR
* No diagnosis of hypertension in the past year but did have the last office blood pressure ≥140 mm Hg systolic or ≥90 mmHg diastolic

Exclusion Criteria:

* Persistent atrial fibrillation as indicated in the electronic health record (EHR)
* Stage IV or more severe kidney disease, defined as estimated glomerular filtration rate <30 per 1.73 m2 or currently on renal replacement therapy (i.e. hemodialysis or peritoneal dialysis)
* Diagnosis of dementia as indicated in the electronic health record

Ages: 65 Years to 85 Years | Sex: All
Age Groups: Older Adult
Study Population: This study will take place in several Northwestern Medicine Group outpatient primary care clinic settings. Patients at these practices will be eligible for inclusion in the primary study population if they have diagnosed hypertension, are 65 to 85 years old, have Medicare insurance, and have their last two prior office blood pressures ≥140 mm Hg systolic or ≥90 mm Hg diastolic. Patients at these practices will be eligible for inclusion in the secondary study population if either they meet the inclusion criteria for the primary population or they are 65 to 85 years old, have Medicare insurance and either have diagnosed hypertension but do not have their last two office blood pressures prior ≥140 mm Hg systolic or ≥90 mm Hg diastolic, or they do not have hypertension diagnosed and have their most recent prior office blood pressure ≥140 mm Hg systolic or ≥90 mm Hg diastolic.
Sampling Method: Non-Probability Sample
Enrollment: 17290 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-08-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Performance measure Controlling High Blood Pressure (NQF 0018) | 6 months
  Proportion of eligible hypertension patients with most recent eligible blood pressure in the measurement period <140/90 mm Hg, binary
Performance measure Controlling High Blood Pressure (NQF 0018) | 3 months
  Proportion of eligible hypertension patients with most recent eligible blood pressure in the measurement period <140/90 mm Hg, binary

SECONDARY OUTCOMES:
Systolic blood pressure at the most recent office visit | 6 months
  Systolic blood pressure at the most recent office visit (mm Hg), continuous
Systolic blood pressure at the most recent office visit | 3 months
  Systolic blood pressure at the most recent office visit (mm Hg), continuous
Antihypertensive medication intensification | 6 months
  Antihypertensive medication intensification, count
Antihypertensive medication intensification | 3 months
  Antihypertensive medication intensification, count
Systolic blood pressure measured by home readings | 6 months
  Systolic blood pressure measured by home (mm Hg) measured using RPM, continuous
Systolic blood pressure measured by home readings | 3 months
  Systolic blood pressure measured by home (mm Hg) measured using RPM, continuous
Remote patient monitoring intensity | 6 months
  Number of RPM BP measurements in months during which any BP measurement was performed, count
Remote patient monitoring intensity | 3 months
  Number of RPM BP measurements in months during which any BP measurement was performed, count
RPM use | 6 months
  Any remote BP transmitted, binary
RPM use | 3 months
  Any remote BP transmitted, binary
RPM BP monitoring uptake | up to 6 months
  Time from BP RPM prescription to first BP RPM measurement, time-to-event
RPM BP monitoring discontinuation | up to 6 months
  Time from first BP RPM measurement until end of first 30-day period with no RPM BP readings, time-to-event
Controlling high blood pressure--office only | 6 months
  Proportion of eligible hypertension patients with most recent eligible office blood pressure in the measurement period <140/90 mm Hg, binary
Controlling high blood pressure--office only | 3 months
  Proportion of eligible hypertension patients with most recent eligible office blood pressure in the measurement period <140/90 mm Hg, binary

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Persell, MD, MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Persell SD, Petito LC, Anthony L, Peprah Y, Lee JY, Campanella T, Campbell J, Pigott K, Kadric J, Duax CJ, Li J, Sato H. Prospective Cohort Study of Remote Patient Monitoring with and without Care Coordination for Hypertension in Primary Care. Appl Clin Inform. 2023 May;14(3):428-438. doi: 10.1055/a-2057-7277. Epub 2023 Mar 18. PMID 36933552